CLINICAL TRIAL: NCT00450710
Title: Phase IV Study of Neuroendocrine Brake Surgical Procedure for Type 2 Diabetes Mellitus
Brief Title: Neuroendocrine Brake for Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AS06005
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Procedure: ileal interposition with a sleeve gastrectomy

SUMMARY:
Evaluation to determine the safety of two laparoscopic procedures to control T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. - Male and female between 18 and 65 years.
2. BMI 25.1 - 34.9.
3. Type 2 diabetic patients on oral anti-diabetic agents and/or insulin treatment for a minimum of 12 months prior the enrollment.
4. Diagnosis of T2DM for at least 3 years.
5. Patient has been under routine care of hte study physician or another physician that can supply a reliable medical record for at least 3 years.
6. HbA1c >/ 7.5 documented for at least 3 months.
7. Stable weight (nor significant weight change (>3%) over the 3 months prior to enrollment.
8. Stable medication for at least one month prior to enrollment except for diabetes medications which should be stable for at least 3 months prior to enrollment.
9. Ability and willingness to return for all scheduled visits and participate in recommended parameter setting and physician recommended medical/laboratory assessments.

Exclusion Criteria:

1. Prior abdominal surgery, except laparoscopic cholecystectomy.
2. Taking appetite suppressant.
3. Severe eating disorders.
4. Severe pulmonary, renal or cardiac disease.
5. Obese due to a clinically diagnosed endocrine disorder.
6. Subjects with impaired liver function.
7. History of peptic ulcer disease.
8. History of malignant disease.
9. Use of prescription, over the counter or herbal weight loss products.
10. Pregnant or planning on pregnancy while enrolled in study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-03; Primary Completion 2008-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and efficacy of the ileal interposition associated with a sleeve gastrectomy and the ileal interposition associated with a diverted sleeve gastrectomy.

SECONDARY OUTCOMES:
Evaluate neurohormonal effect in treating T2DM.
Improvement or control of blood glucose levels.
Improvement or control of comorbidities associated with T2DM.
Hormonal effect and effect of the operations on diabetes related and total mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Noreen A Gannon, Study Director — Medtronic - MITG; Aureo DePaula, MD, Principal Investigator — Hospital de Especialidades
Locations (1):
- Hospital de Especialidades, Goiânia, Brazil